CLINICAL TRIAL: NCT00004731
Title: Effects of Coenzyme Q10 in Early Parkinson's Disease
Brief Title: Parkinson's Disease Treatment With Coenzyme Q10
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01NS036714 (NIH)
Record Dates: First submitted 2000-02-25; First posted 2000-02-28 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; coenzyme Q10
MeSH Terms: conditions — Parkinson Disease | interventions — coenzyme Q10

INTERVENTIONS:
Drug: Coenzyme Q10

SUMMARY:
The purpose of this study is to compare the effects of varying dosage of coenzyme Q10 (CoQ10) versus a placebo in the treatment of Parkinson's disease (PD) in patients with early, untreated PD.

DETAILED DESCRIPTION:
Four groups of 20 subjects/group of subjects will be randomly assigned to receive CoQ10 (at doses of 300, 600 or 1200 mg/day) or matching placebo. A subject must have early PD that does not require treatment. A subject will be evaluated at a Screening Visit, a Baseline Visit (after which the subject begins to take the study drug) and visits at 1, 4, 8, 12, and 16 months after the baseline visit. The subject will be followed until she/he needs treatment with levodopa or for a maximum of 16 months. Because CoQ10 is a component of the mitochondria (the part of a cell that makes energy), blood samples will be taken at the baseline visit and the last visit to study mitochondrial function.

ELIGIBILITY:
Inclusion Criteria:

* The subjects must have the three cardinal features of PD: slowness of movement, resting tremor and rigidity. The signs of PD must be greater on one side.

Exclusion Criteria:

* Disorders that mimic PD.
* Other serious medical problems.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-09; Study Completion 2003-10

CONTACTS AND LOCATIONS:
Overall Officials: Clifford W. Shults, M.D., Principal Investigator — University of California, San Diego
Locations (1):
- University of Rochester, Rochester, New York, United States